CLINICAL TRIAL: NCT04259827
Title: On-line Cognitive Training for Mild Cognitive Impairment in Parkinson's Disease: a Randomized Single-blind Study Using Wearing Sensors Technology
Brief Title: On-line Cognitive Training for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Pilotto, Neurology Department Director, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/01
Record Dates: First submitted 2020-01-18; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study is a 3-arms single-blind parallel study. The patients are not blind to treatment , the investigators who will perform the baseline and follow-up assessment will be blinded to the treatment performed.
Who Masked: Investigator
Masking Description: The cognitive, motor and wearing sensors assessment will be performed by investigators blind to the treatment performed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online cognitive training (Experimental): 6-week online personalized cognitive training using Neuronation platform 4 training session three times a week. Each session is composed of 5 exercises from one out of 4 cognitive domains: Memory, Attention, Speed and Reasoning
  Interventions: Other: Neuronation
- Aspecific online games (Active Comparator): online application not created with a cognitive training purpose, for the same amount of time and frequence as the experimental group
  Interventions: Other: Aspecific online games
- No online cognitive training (No Intervention): normal clinical follow-up without cognitive training or gaming

INTERVENTIONS:
Other: Neuronation — Online cognitive training app, with exercises created for patients with mild cognitive impairment
  Arms: Online cognitive training
Other: Aspecific online games — Online gaming without cognitive training
  Arms: Aspecific online games

SUMMARY:
Application of online cognitive training in patients affected by Parkinson's disease and mild cognitive impairment. The treatment consists of a 6-week on-line cognitive training preceded and followed by neurological, neuropsychological and motor assessment.

DETAILED DESCRIPTION:
At the recruitment, participants will undergo a neurological visit, a neuropsychology assessment (2 tests for each considered cognitive domain: memory, attention, visuospatial, executive function, language) and a motor assessment with wearing sensors under supervised conditions.

In the treatment arm only, patients will have the Neuronation application installed on their personal technology device (smartphone or tablet) and are asked to complete 4 training session three times a week. Each session is composed of 5 exercises from one out of 4 cognitive domains: Memory, Attention, Speed and Reasoning. The training is tailor made, the complexity of the exercises is adjusted online, based on the patient's performance.

Participants are re-assessed at the end of the 6-week cognitive training (T1) to find out its effects on cognition and motor ability. The same assessment is administered also after 1 (T2) and 3 (T3) months from the end of the cognitive training to test long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Ease of use of at home internet connection
* Active presence of a caregiver to help with the use of the App
* Sufficient physical ability to use a technological device
* Signature of informed consent

Exclusion Criteria:

* Presence of systemic pathologies potentially responsible for cognitive deficits
* Presence of pathologies of the Central Nervous system potentially associated with cognitive deficits
* No access to internet connection
* Cognitive rehabilitation within the previous 6 months
* Major depression (assessed by Beck Depression Inventory at baseline)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-02-10 (Estimated)

PRIMARY OUTCOMES:
Trial making B performance, total score (0-240 seconds) | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Trial making B performance, total score (0-240 seconds)
Sum of total Z-score of cognitive assessment (-30 to 30) | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Sum of total Z-score of cognitive assessment (-30 to 30)
Supervised gait performance normal gait | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Step variability using wearing sensors technology in one-minute supervised walking
Supervised gait performance dual task gait | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Step variability using wearing sensors technology in one-minute supervised dual task walking
Parkinson´s disease Quality of life questionnire (PDQ-39) (0-117 points) | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  PDQ-39 will be assessed in patients
Quality of life - caregivers | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Caregiver Burden will be assessed with Dyadic relationship scale

SECONDARY OUTCOMES:
Unified parkinson´s disease Rating Scale part 3 (0-132 points) | Changes between baseline, immediately after the end of intervention, after 1 month and 3 monthss
  Total Movement Disorder Society-Unified Parkinson's disease Rating Scale part 3 motor score
Instability measures | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Wearing sensors-based instability assessment (area of sway)
Turning performances | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Wearing sensors based turning speed in timed up and go test
Dual task performance in circular walking (0-240 seconds) | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Time performed in dual-task circular walking
Short Physical performance battery (SPPB), total time (0- 60 seconds) | Changes between baseline, immediately after the end of intervention, after 1 month and 3 months
  Short Physical performance battery

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Padovani, Prof, Principal Investigator — Università degli Studi di Brescia
Locations (2):
- Italy (2):
  - Department of Neurology ASST Spedali Civili Brescia, Brescia, Lombardy
  - Parkinson's disease Rehabilitation Centre, Trescore Balneario, Lombardy

IPD SHARING:
Plan to Share IPD: Yes
Wearing sensors data will be available after completion of the trial.
Supporting Information: Study Protocol, SAP
Time Frame: After the completion of the trial
Access Criteria: upon reasonable request